CLINICAL TRIAL: NCT06432140
Title: An Open, Dose-escalating and Dose Confirmation Trial to Evaluate the Safety and Efficacy of VGN-R09b by Intra Putamen Injection in Patients With Severe Aromatic L-amino Acid Decarboxylase (AADC) Deficiency
Brief Title: A Trial to Evaluate Safety and Efficacy of a Product Named VGN-R09b in Severe AADC Deficiency
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Vitalgen BioPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGN-R09b-102
Record Dates: First submitted 2024-05-17; First posted 2024-05-29 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Aromatic L-amino Acid Decarboxylase Deficiency
Keywords: AADC; AAV9; Central Nervous System (CNS) gene therapy
MeSH Terms: conditions — Aromatic amino acid decarboxylase deficiency

STUDY DESIGN:
Intervention Model Description: VGN-R09b will be injected into bilateral putamen by stereotactic surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VGN-R09b injection (Experimental): Different levels of VGN-R09b will be injected into bilateral putamen by stereotactic surgery
  Interventions: Genetic: VGN-R09b injection

INTERVENTIONS:
Genetic: VGN-R09b injection — Two levels of VGN-R09b will be injected into bilateral putamen in dose-escalating phase, and one dose level will be injected in dose confirming phase

SUMMARY:
This trial includes dose-escalating part (phase 1) and dose confirming part, to prove the safety and efficacy of VGN-R09b to treat patients with severe AADC deficiency

DETAILED DESCRIPTION:
Aromatic L-amino acid decarboxylase (AADC) is an enzyme responsible for the final step in the synthesis of neurotransmitters dopamine and serotonin. AADC deficiency is a rare genetic disorder. VGN-R09b is a kind of Gene therapy with adeno-associated virus (AAV) serotype 9 (AAV9) driven human AADC (hAADC) being injected directly into putamen.

This is an open, dose-escalating and dose confirming study. The sponsor plans to explore two dose levels (6.0×1011vg and 1.28×1012vg) in dose-escalating phase (three subjects each cohort), then plans to have 10 subjects enrolled for dose confirmation phase.

This study is to give evidence for the safety and efficacy of VGN-R09b treatment for patients with severe Aromatic L-amino acid decarboxylase (AADC) deficiency.

ELIGIBILITY:
Inclusion Criteria:

1. The child patient has to be ≥18 months old and < 8 years old, and a head circumference big enough for surgery as judged by investigator.
2. Historical diagnosis of AADC deficiency with clinical symptoms consistency, AND with Molecular genetic confirmation of homozygous or compound heterozygous mutation point of IVS6+4A>T in DDC gene.
3. With Plasma AADC activity less than or equal to 12 pmol/min/mL.
4. Motor development at baseline <3 months (head fully uncontrollable at baseline）, and Failed to benefit from standard medical therapy (dopamine agonists, monoamine oxidase inhibitor or related form of Vitamin B6) at discretion of investigators.
5. Parent(s)/legal guardian(s) with custody of subject must give their consent for subject to enroll in the study.
6. Parent(s)/legal guardian(s) of the subject must agree to comply with the requirements of the study, including providing disease information and support disease assessment of symptoms.

Exclusion Criteria:

1. Intracranial neoplasm or any structural brain abnormality or lesion (e.g., severe brain atrophy, white matter degenerative changes), which, in the opinion of the study investigators, would confer excessive risk and/or inadequate potential for benefit.
2. Presence of other significant medical or neurological conditions that would create an unacceptable operative or anesthetic risk (including congenital heart disease, respiratory disease with home oxygen requirement, history of serious anesthesia complications during previous elective procedures, history of cardiorespiratory arrest), liver or renal failure, malignancy, or HIV positive.
3. Severe coagulopathy, or need for ongoing anticoagulant therapy.
4. clinically active infection or with severe infection within 12 weeks before screening (e.g. adenovirus or herpes virus, pneumonia, sepsis, central nervous system infection).
5. Previous stereotactic neurosurgery, or any gene/cell therapy.
6. Received live vaccination within 4 weeks.
7. Contraindication to sedation during surgery or imaging studies (PET or MRI).

Ages: 18 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs), Serious Adverse Events (SAEs) | up to Week 52
  Vital signs, physical examination, laboratory test will be monitored after drug injection
Number of subjects who achieved motor development milestones | up to 24 months
  Four milestones, including Head control, Sit independently, Stand/stepping with support, Walk with minimal assistant, would be assessed according to definition in Peabody Developmental Motor Scale 2nd edition (PDMS-2). Each milestone would be scored as 0, 1 or 2, and score 2 means achievement of the milestone.

SECONDARY OUTCOMES:
Change in brain AADC activity | up to 5 Years
  Increase in signal in the putamen and nigra on Fluorodopa-PET imaging as brain AADC activity measure
Change in Cerebrospinal Fluid (CSF) neurotransmitter metabolite concentrations | up to 5 Years
  Neurotransmitter metabolite concentrations of Homovanillic Acid/Hydroxyindoleacetic Acid (HVA/5-HIAA) would be measured
Change from baseline in motor function | up to 5 Years
  Motor function would be assessed by Peabody Developmental Motor Scale 2nd edition (PDMS-2). The score ranges from 0 to 482, and higher score means the better in motor function.
Change in number of Clinical symptoms | up to 5 Years
  Number of disease related symptoms
Viral shedding | up to 1 week
  Concentrations of Viral genome in serum/urine would be measured
Immunogenicity after injection | up to 26 weeks
  Subject number with positive antibodies of AAV9/AADC/Glial Cell Line-Derived Neurotrophic Factor (GDNF) in blood would be reported
Number of Adverse Events (AEs), Serious Adverse Events (SAEs) in Long-term follow-up | up to 5 Years
  Drug-related AEs and SAEs would be monitored as long as 5 years after injection

CONTACTS AND LOCATIONS:
Overall Officials: Xiumin Wang, MD, Principal Investigator — Shanghai Children's Medical Center, affiliated to Shanghai Jiao Tong University School of Medicine